CLINICAL TRIAL: NCT02910414
Title: A Pivotal, Multicenter, Blinded, Sham Procedure-Controlled Trial of Renal Denervation by the Peregrine System™ Kit, in Subjects With Hypertension
Brief Title: TARGET BP I Clinical Trial
Acronym: TARGET BP I
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ablative Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR0002
Record Dates: First submitted 2016-09-16; First posted 2016-09-22 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
Keywords: Renal Denervation; Alcohol
MeSH Terms: conditions — Hypertension | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Treated with Peregrine System Kit (Experimental): The experimental group will receive an infusion of Dehydrated Alcohol Injection, USP into the perivascular space of the renal arteries with the Peregrine Catheter. A total of 0.6mL of the alcohol will be delivered to the perivascular space of each renal artery. The drug will only be delivered once to each renal artery during the treatment procedure.
  Interventions: Drug: Dehydrated alcohol
- Renal Angiography Only (Sham Procedure) (Sham Comparator): The sham control group will only have diagnostic renal angiography performed. There will be no insertion of the Peregrine Catheter and no alcohol infusion (i.e. no renal denervation).
  Interventions: Device: Peregrine System Kit (Sham Procedure)

INTERVENTIONS:
Drug: Dehydrated alcohol — Dehydrated Alcohol Injection, USP is used in the study.
  Other Names: Ethanol
  Arms: Treated with Peregrine System Kit
Device: Peregrine System Kit (Sham Procedure) — Pre-procedural diagnostic renal angiography only, performed for confirmation of anatomical eligibility prior to randomization
  Arms: Renal Angiography Only (Sham Procedure)

SUMMARY:
The TARGET BP I Trial is a randomized, blinded, multi-center, international, sham-procedure controlled trial, comparing renal denervation performed with the Peregrine System Kit in the treatment group to the sham control group (without renal denervation - no alcohol infusion). Subjects will be randomized in a 1:1 fashion to treatment versus sham control via central randomization.

DETAILED DESCRIPTION:
The TARGET BP I Trial is a randomized, blinded, multi-center, international, sham-procedure controlled trial, comparing renal denervation performed with the Peregrine System Kit in the treatment group to the sham control group (without renal denervation - no alcohol infusion). Subjects will be randomized in a 1:1 fashion to treatment versus sham control via central randomization.

The TARGET BP I clinical trial uses a percutaneous catheter to deliver very small amounts of alcohol (neurolytic agent). The patient population for this trial is comparable to those used in other renal denervation studies, but also incorporates lessons learned from recent trials of renal denervation. This is to enable the study of an optimized patient population who stands to benefit from the intervention, in a manner that reduces possible study bias.

This trial is intended to evaluate the safety and efficacy of the Peregrine Catheter when used to deliver a 0.6 mL volume of alcohol to the perivascular area of the respective renal arteries while patients are adequately managed with oral antihypertensive medications.

ELIGIBILITY:
Inclusion Criteria:

1. Has 3 office blood pressure measurements with a mean office systolic blood pressure (SBP) of ≥150 mmHg and ≤180 mmHg, AND a mean office diastolic blood pressure (DBP) of ≥90 mmHg when receiving 2 to 5 antihypertensive medications.
2. Has a mean 24-hour ambulatory SBP of ≥135 mmHg and ≤170 mmHg with ≥70% valid readings

Exclusion Criteria:

1. Subject has renal artery anatomy abnormalities.
2. Subject has an estimated glomerular filtration rate (eGFR) of ≤45 mL/min/1.73 m2, based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation; or is on chronic renal replacement therapy.
3. Subject has documented sleep apnea.
4. Subject has any of the following conditions: severe cardiac valve stenosis, heart failure (New York Heart Association [NYHA] Class III or IV), chronic atrial fibrillation, and known primary pulmonary hypertension (>60 mmHg pulmonary artery or right ventricular systolic pressure).
5. Subject is pregnant or lactating at the time of enrollment or planning to become pregnant during the trial time period (female subjects only).
6. Subject is being treated chronically (e.g. daily use) with NSAIDs, immunosuppressive medications, or immunosuppressive doses of steroids. Aspirin therapy and nasal pulmonary inhalants are allowed.
7. Subject has a history of myocardial infarction, unstable angina pectoris, or stroke/TIA within 6 months prior to the planned procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in mean systolic ABPM | 3 months
  The change in mean 24-hour ambulatory SBP from baseline to 3 months post-procedure

SECONDARY OUTCOMES:
Proportion of subjects with major adverse events | 30 days
  Major Adverse Events as defined in the clinical protocol
Major Adverse Events | 3, 6, and 12 months and 2 and 3 years
  Major Adverse Events as defined in the clinical protocol
Decrease in eGFR > 25% | 3 and 6 months
  Decrease in eGFR > 25% at 3 and 6 months
Changes in eGFR | 3 and 6 months
  Changes in eGFR at 3 and 6 months
Adverse event rate | Procedure date, discharge date (an average of 1 day), 5-day, 4 weeks, 8 weeks, 3 months, 4 months, 5 months, 6 months, 1 year, 2 years and 3 years
  Adverse event rate at procedure, discharge, and at all follow-up visits
Device success | Procedure date (day 0)
  Device success, defined as successful introduction of the catheter, navigation to the treatment site, deployment of the needles, and infusion of the alcohol to the intended area via the Peregrine Catheter as intended for use
Procedure success | Hospital discharge date (an average of 1 day)
  Procedure success defined as device success and freedom from serious adverse events related to the product or the procedure, during the procedure and prior to hospital discharge from the index procedure.
Change of office systolic blood pressure | 8 weeks
  Change of office systolic blood pressure from baseline to 8 weeks
Change of diastolic office blood pressure | 3 and 6 months
  Change of diastolic office blood pressure from baseline to 3 and 6 months
Change of 24-hour mean diastolic ABPM | 3 and 6 months
  Change of 24-hour mean diastolic ABPM from baseline to 3 and 6 months
Change of 24-hour mean systolic ABPM | 6 months
  Change of 24-hour mean systolic ABPM from baseline to 6 months
Changes in antihypertensive regimen | 3 months
  Changes in antihypertensive regimen from procedure to 3 months post-procedure
ABPM responders (5 mmHg) | 3 months
  ABPM Responders, defined as the proportion of subjects with a drop of ≥5 mmHg in 24-hour ambulatory SBP at 3 months compared with baseline.
Office BP responders (10 mmHg) | 3 months
  Office BP Responders, defined as the proportion of subjects with a drop of ≥10 mmHg in office SBP at 3 months compared with baseline.
Change in mean office SBP | 6 months
  Change in mean office SBP from baseline to 6 months post-procedure
Change in mean daytime ambulatory SBP | 3 months
  Change in mean daytime ambulatory SBP from baseline to 3 months post procedure.
Change in mean daytime ambulatory SBP | 6 months
  Change in mean daytime ambulatory SBP from baseline to 6 months post procedure.
Change in mean daytime ambulatory DBP | 3 and 6 months
  Change in mean daytime ambulatory DBP from baseline to 3 months and then 6 months post procedure.
Changes (decreases or increases) in antihypertensive medication regimen from 3 months to 6 months post-procedure | 3 and 6 months
  Changes (decreases or increases) in antihypertensive medication regimen from 3 months to 6 months post-procedure (titrated according to standardized formula to maintain a target office SBP of < 140 mmHg and ≥ 90 mmHg).
Changes (decreases or increases) in antihypertensive medication regimen from procedure to 6 months post-procedure | 6 months
  Changes (decreases or increases) in antihypertensive medication regimen from procedure to 6 months post-procedure (titrated according to standardized formula to maintain a target office SBP of <140 mmHg and ≥90 mmHg)
Change in mean nighttime ambulatory SBP | 3 and 6 months
  Change in mean nighttime ambulatory SBP from baseline to 3 months and then 6 months post procedure.
Change in mean nighttime ambulatory DBP | 3 and 6 months
  Change in mean nighttime ambulatory DBP from baseline to 3 months and then 6 months post procedure.
Reduction of office SBP and DBP to normal | 3, 6, and 12 months
  Reduction of office SBP and DBP to normal (<140/90 mmHg) at 3, 6 and 12 months as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Piedmont Heart Institute; Michael Weber, MD, Principal Investigator — SUNY Downstate Medical; Atul Pathak, MD, Principal Investigator — Clinique Pasteur; Felix Mahfoud, MD, Principal Investigator — Klinik fur Innere Medizin III
Locations (5):
- United States (5):
  - Cardiology PC, Birmingham, Alabama
  - Piedmont Heart Institute, Atlanta, Georgia
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kandzari DE, Weber MA, Pathak A, Zidar JP, Saxena M, David SW, Schmieder RE, Janas AJ, Langer C, Persu A, Mendelsohn FO, Ameloot K, Foster M 3rd, Fischell TA, Parise H, Mahfoud F. Effect of Alcohol-Mediated Renal Denervation on Blood Pressure in the Presence of Antihypertensive Medications: Primary Results From the TARGET BP I Randomized Clinical Trial. Circulation. 2024 Jun 11;149(24):1875-1884. doi: 10.1161/CIRCULATIONAHA.124.069291. Epub 2024 Apr 8. PMID 38587557
- [Derived] Bertog S, Sharma A, Mahfoud F, Pathak A, Schmieder RE, Sievert K, Papademetriou V, Weber MA, Haratani N, Lobo MD, Saxena M, Kandzari DE, Fischell TA, Sievert H. Alcohol-Mediated Renal Sympathetic Neurolysis for the Treatment of Hypertension: The Peregrine Infusion Catheter. Cardiovasc Revasc Med. 2021 Mar;24:77-86. doi: 10.1016/j.carrev.2020.09.003. Epub 2020 Sep 7. PMID 32958438